CLINICAL TRIAL: NCT07362875
Title: Development of Quantitative Muscle Imaging as a Biomarker of Disease Endpoints in Myotonic Dystrophy (DeQoDE-DM)
Brief Title: Development of Quantitative Muscle Imaging as a Biomarker of Disease Endpoints in Myotonic Dystrophy
Acronym: DeQoDE-DM
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00125282
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Myotonic Dystrophy
Keywords: dystrophia myotonica; muscular dystrophy; skeletal myopathy
MeSH Terms: conditions — Myotonic Dystrophy; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A subset of 20 subjects with DM (approximately 10 subjects with DM1 and 10 subjects with DM2) and 5 controls will undergo needle muscle biopsies (tibialis anterior for DM1 and controls, vastus lateralis for DM2) after completion of the MRI scan and Coarctation of the Aorta (COAs). These subjects will sign a separate consent form for muscle biopsy sub-study. The biopsy procedure will involve 3 study visits: screening, biopsy, and follow-up visits. Depending on the availability of the subjects, research staff, and facilities, it is possible that the screening and biopsy visits can be combined into one visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM subjects: 1. Age 18 - 65 years
  2. Diagnosis of DM1 or DM2 by clinical or genetic criteria. If DM1 or DM2 was diagnosed by clinical criteria, a first-degree relative must have genetic testing confirmation and sign a genetic consent form to release their genetic information.
  3. Clinically affected, as defined by muscle weakness or myotonia
  4. Ambulate independently (a walker is not permitted)
  5. Able to provide informed consent for participation in the study
- Control subjects: 1. Age 18 - 65 years old
  2. Healthy as defined by no significant medical or neurological conditions
  3. Able to provide informed consent for participation in the study

SUMMARY:
Myotonic dystrophy (dystrophia myotonica; DM), the most prevalent form of muscular dystrophy in adults, is characterized by progressive myopathy, myotonia, and multi-systemic involvement. DM causes severe disability and profoundly affects the patient's quality of life. Currently, no effective treatments are available that alter the course of the disease, but ongoing clinical trials are underway.

DETAILED DESCRIPTION:
Past and current clinical trials in DM1 have relied on muscle biopsies to evaluate pathology and measure drug activity. However, this method is invasive and inefficient for long-term monitoring. What is lacking are non-invasive imaging biomarkers capable of providing comparable data, which would enhance trial planning, accelerating drug development while reducing morbidity and costs. Non-invasive muscle imaging, particularly through Quantitative Magnetic Resonance Imaging (qMRI), is essential to better understand how DM affects muscle structure. Moreover, the relationships between Magnetic Resonance Imaging (MRI) measures, disease severity, and Ribonucleic Acid (RNA) splicing outcomes from muscle tissues in the same DM patients are not yet known. As MRI has been relatively unstudied in DM, there needs to be a comprehensive baseline characterization of muscle structure and its relationship to clinical endpoints and RNA-associated disease processes. This will help evaluate the potential of qMRI as a biomarker of disease severity in DM.

ELIGIBILITY:
Inclusion Criteria:

DM subjects

* Age 18 - 65 years
* Diagnosis of DM1 or DM2 by clinical or genetic criteria. If DM1 or DM2 was diagnosed by clinical criteria, a first-degree relative must have genetic testing confirmation and sign a genetic consent form to release their genetic information
* Clinically affected, as defined by muscle weakness or myotonia
* Ambulate independently (a walker is not permitted)
* Able to provide informed consent for participation in the study

Control subjects

* Age 18 - 65 years old
* Healthy as defined by no significant medical or neurological conditions
* Able to provide informed consent for participation in the study

Exclusion Criteria:

* Cardiac pacemaker, defibrillator, metal implants, or other contraindications for MRI
* Use of anabolic or catabolic agents within one year of entry
* History of lumbar spine or leg surgery, lumbar radiculopathy, or peripheral neuropathy
* BMI > 35 because obesity compromises positioning on the MR scanner
* Pregnancy
* For muscle biopsy, history of bleeding disorders or on anticoagulation. Subjects taking nonsteroidal anti- inflammatory agents will be asked to discontinue these medications 7 days prior to muscle biopsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The selection criteria will minimize the heterogeneity effects and mirror DM subjects likely to be selected for clinical trials, who are typically mildly to moderately affected. Subjects will be recruited from the Wake Forest Neuromuscular Clinic and nearby medical centers (Duke University, UNC Chapel Hill, and Atrium Health in Charlotte).
  Since DM2 is rarer than DM1 and patients live across the country, additional recruitment efforts will target DM2 subjects through the Myotonic Dystrophy Foundation Family Registry (MDFR).
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Contractile muscle volume (CMV, cm3) | Baseline
  Contractile muscle volume (CMV, cm3) of individual muscles and the total CMV within the thigh (anterior, medial, posterior) and calf (anterior, lateral, posterior) compartments
Muscle fat fraction (MFF, %) | Baseline
  Muscle fat fraction (MFF, %) of individual muscles and the total CMV within the thigh (anterior, medial, posterior) and calf (anterior, lateral, posterior) compartments

SECONDARY OUTCOMES:
Average measures of Manual muscle testing (MMT) | Baseline
  MMT will be performed in 7 different muscle groups (hip flexors, hip abductors, knee flexors, knee extensors, ankle dorsiflexors, plantar flexors, and neck flexor) in standardized positions. Each group will be scored using a 13-point modified Medical Research Council (MRC) scale and standardized positions. Where 0 is paralysis, 1 is a flicker/trace contraction, 2 is movement with gravity eliminated, 3 is movement against gravity, 4 is movement against some resistance, and 5 is normal strength against full resistance - higher scores denoting stronger muscles
Average measures of Quantitative Muscle Testing (QMT) | Baseline
  QMT of the leg muscles (hip flexors, hip abductors, knee extensors, knee flexors, ankle dorsiflexors, and plantar flexors) will be performed using a hand-held dynamometer in standardized positions. During the measurement, the subject will be instructed to increase to maximum exertion over a few seconds without jerking, and to maintain this effort until the evaluator give the command to relax (3-5 seconds). The clinical evaluator will hold the dynamometer stable, and the subject will be asked to push as hard as possible against the applicator, but with a slow build-up of force. The subject will perform each push three times with up to a 30-second pause between each trial. The average and highest scores obtained will be used for analysis.
Average measures of grip strength (pounds or kilograms) | Baseline
  Use Jamar handgrip dynamometer to test handgrip strength. We will test each subject three trials, starting with a dominant hand first, then a non-dominant hand. An average score in each hand will be used for analysis. Higher scores denote stronger grip strength - It works by squeezing the device to its maximum, revealing strength in pounds or kilograms (up to 200 lbs/90 kg)
Average measures of pinch strength | Baseline
  The subject will perform quantitative pinch strength testing with a pinch gauge - higher numbers denote stronger pinch strength - Normal range: 10-20 pounds of force
The 6-minute walk test (6MWT) times | Baseline
  walking ability in muscular dystrophies, the 6MWT probably offers the best combination of reliability, sensitivity, clinical significance, and feasibility for clinical trials. The procedures will be performed in a standardized manner following the guidelines of the American Thoracic Society. Lower times denote faster walks
gait speed times | Baseline
  Subjects will be instructed to walk at maximum speed in a long corridor with an even surface over 10 meters with a still-standing start and a "flying" finish. The subjects will be instructed to continue walking to a target 2.5 meters beyond the mark at 4 and 10 meters, where the clinical evaluator stands. The time will be measured with the stopwatch and is started on the word "Go" ("Ready-Set-Go") until subject reaches a 4 and 10-meter mark. Lower times denotes faster speeds
step test amount | Baseline
  The subject will stand unsupported 5 cm in front of a block (maximum height 10 cm) and make as many "full steps" as possible during 15-second period. One step comprises placing one foot fully up onto and then down off the block. Both legs will be tested, one foot at a time. The subject will allow some practice steps and then one test attempt per leg. If balance is lost during the trial, the completed steps will be reported. Clinical Evaluator will kneel by the block and holds it to ensure it remains steady during the test. higher scores denotes better balance and strength
sit-to-stand test amount | Baseline
  The test will be administered using a standard chair with a seat height of 17 inches (43.2 cm) and rubber tips on the legs. The test begins with the subject seated in the middle of the chair, back straight, feet approximately shoulder-width apart and place on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance when standing. Arms are crossed and held against the chest. At the signal "go," the subject will rise to a full stand and then return to the initial seated position. The subjects will be encouraged to complete as many full stands as possible within a 30-second time limit. The score will be the total number of stands executed correctly. Incorrectly executed stands will not be counted - higher scores denotes better balance and strength
Short Physical Performance Battery (SPPB) Scores | Baseline
  The physical performance will be assessed using the expanded SPPB commonly used in research. The SPPB measures physical function using three components: 4-meter natural gait speed, time to complete five chair rises, and standing balance with a narrow base of support. Each component is scored on a 0-4 scale and summed for an overall score range of 0-12. The SPPB is a reliable and validated measure of physical function in the older population that can be collected safely and easily at clinic, home, or hospital setting. Overall scores and components of SPPB are highly predictive of clinical outcomes, including disability, hospitalization, and death. The SPPB is also sensitive to change over time and responsive to exercise training. A clinically meaningful but small change in SPPB score is 0.5 units, and a substantial change is 1.0 units
Nine-Hole Peg Test (9HPT) times | Baseline
  The test will evaluate upper extremity function, specifically fine dexterity, and coordination. test each subject once, starting with a dominant hand first, then a non-dominant hand. One practice trial (per hand) should be provided before timing the test. The subjects will be instructed to pick up the pegs one at a time using one hand only and put them into the holes one at a time and return each of them to the container. Lower times denotes higher dexterity and coordination
Time Up and Go (TUG) times | Baseline
  TUG is used to evaluate various aspects of dynamic stability related with falls. A TUG time > 14 seconds is associated with falls in DM1. The TUG includes rising from a chair, walking 3 meters, turning, walking back, and sitting down. The TUG shows good test-retest reliability (ICC > 0.8) in individuals with DM1 - scores under 10 seconds are normal, under 20 seconds indicate good mobility, while over 30 seconds suggests significant impairment, requiring assistance and indicating a high fall risk, with 14+ seconds signaling increased risk.
DM1-Activity and Participation Scale (DM1-Activ) Scores | Baseline
  The DM1-Activ is a 25-item instrument, designed to assess activity limitations in individuals with DM1. It has been validated as a disease-specific PRO measure for assessing activity limitations in DM1 with good internal consistency and constructive validity. It captures the impact of DM1 on daily activities and physical function, making it a valuable tool for clinical trials and disease monitoring - using response options from "impossible" to "without difficulty"
Patient-Reported Outcomes Measurement Information System (PROMIS-10) Scores | Baseline
  assessing global health (physical and mental) and social well-being. It evaluates health symptoms and quality of life sub-domains such as pain, fatigue, physical activity, and global health (GH). PROMIS is well-validated with chronic neurological conditions, demonstrating strong internal consistency and cross-sectional validity. use PROMIS-10, a 10-item questionnaire, assessing multiple health domains. This tool provides less ceiling effect and has been accepted as a key outcome in the NINDS Common Data Elements. The raw responses (1-5 scale) are converted to these T-scores, allowing for interpretation like scores above 60 being moderately worse than average and below 40 being significantly better.
Brief Pain Inventory (BPI) Scores | Baseline
  The short form BPI is designed to measure the interference pain has with patient daily activities. These scales were selected based on their validity, simplicity, ability to detect change in pain with treatment, patient relevance, reliability, test-retest scores, and their previous use in pain studies of the myotonic dystrophy population - uses 0-10 scales to quantify pain severity (worst, least, average, current) and interference with daily life (mood, activity, sleep, etc.), with higher numbers indicating worse pain or interference
Checklist Individual Strength (CIS-fatigue) Scores | Baseline
  The level of fatigue will be assessed using the CIS 'fatigue severity' subscale. It measures the experience of fatigue-associated problems during the past 2 weeks. The CIS-fatigue severity subscale contains eight items (items 1, 4, 6, 9, 12, 14, 16, 20) scored on a 7-point Likert scale. Scores can range between 8 and 56 with higher scores indicating higher levels of fatigue and scores of > 35 or more are indicated severe fatigue
Muscular Impairment Rating Scale (MIRS) Scores | Baseline
  MIRS is a quick, simple, and reliable scale to evaluate muscle impairment in DM1. It has been validated with motor activities and functional status index questionnaire. It is a five-ordinal scale with the definition of the grades as follows: 1=no impairment; 2=minimal signs, as ptosis and nasality, no distal weakness except long finger flexor weakness; 3=distal weakness, no proximal weakness except in elbow extensors; 4=mild to moderate proximal weakness; and 5=severe proximal weakness. This will be tested for DM1 subjects only. The MIRS is useful to monitor severity stages of disease progression and to identify homogeneous groups of patients for trials
presence of edema-liked changes | Baseline
  MRI Short Tau Inversion Recovery (STIR) sequence data will be evaluated for edema-like changes by assessing the presence or absence of signal hyperintensity in each muscle by a consultant radiologist - STIR (Short Tau Inversion Recovery) sequence is a special MRI technique that suppresses (blacks out) the signal from fat, making it excellent for highlighting fluid-filled tissues like edema (swelling), inflammation, tumors, and stress fractures, especially in bone marrow and soft tissues, because it makes these pathologies appear bright against the dark background of fat.

CONTACTS AND LOCATIONS:
Overall Officials: Araya Puwanant, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No